CLINICAL TRIAL: NCT03136796
Title: Alterations of Glycocalyx in Critical Illness and During Major Surgery and Approaches for Glycocalyx Protection
Brief Title: Glycocalyx Damage and Beta-lactam Antibiotics in Surgical Critically Ill
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Vladimir Cerny, Vladimir Cerny, MD, PhD, FCCM, University Hospital Hradec Kralove
Other Study IDs: AZVCR 9307_4
Record Dates: First submitted 2017-04-22; First posted 2017-05-02 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Meropenem; Piperacillin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Meropenem — Patients will receive intravenous antibiotics eighter empirically or based on a culture.
  Other Names: Piperacillin

SUMMARY:
GCX damage and its relationship to pharmacodynamics and pharmacokinetics of beta lactam antibiotics in critically ill Hypothesis to be tested: GCX damage impairs pharmacodynamics and pharmacokinetics of beta-lactam antibiotics in critically ill patients. There is correlation between GCX damage and insufficient beta lactam levels in patients with commonly used dosing. The aim of the study: Evaluation of relationship between GCX damage and pharmacodynamics and pharmacokinetics of beta-lactam antibiotics in critically ill. Type of the study: Observational. Subjects: Adult patients admitted to ICU with beta-lactam antibiotic therapy (meropenem or piperacillin/tazobactam empirically or based on culture results). Sample size calculation: 20 patients (expected correlation coefficient 0,6, alpha error = 0,05) will lead to power study = 0,89. Intervention: none. Data to be recorded and analyzed: Demographics, type of patients (trauma, post surgical, medical, after cardiac arrest), severity score - Apache II, SOFA, fluid balance, a presence of delirium, clinical outcome, sublingual microcirculation by SDF imaging will be recorded three times during antibiotic treatment at the time points for blood samples required for pharmacodynamics and pharmacokinetic analysis, microcirculatory data and Perfused Boundary Region.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to ICU with beta-lactam antibiotic therapy (meropenem or piperacillin/tazobactam empirically or based on culture results).

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to ICU due to sepsis or polytrauma in need for intravenous antibiotic therapy.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Plasmatic concentrations of antibiotics | 6 months
  Concentration of antibiotics will be assessed in plasma after their administration in mmol/l to calculate their pharmacokinetic and pharmacodynamic profile.

SECONDARY OUTCOMES:
Perfused Boundary Region | 6 months
  PBR is a parameter obtained automatically by specialized software after examination of the sublingual microcirculation by handheld microscope that describes the amount of glycocalyx destruction.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Třebeš, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Astapenko D, Jor O, Lehmann C, Cerny V. In situ assessment of the renal microcirculation in mechanically ventilated rats using sidestream dark-field imaging. J Microsc. 2015 Feb;257(2):161-5. doi: 10.1111/jmi.12198. Epub 2014 Dec 24. PMID 25545609
- [Background] Arora N, Islam S, Wafa K, Zhou J, Toguri JT, Cerny V, Lehmann C. Evaluation of iris functional capillary density in experimental local and systemic inflammation. J Microsc. 2017 Apr;266(1):55-59. doi: 10.1111/jmi.12518. Epub 2017 Jan 19. PMID 28102536